CLINICAL TRIAL: NCT05491382
Title: Muscle and Body Temperature Responses During Uphill and Downhill Running
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical malfunctions of key equipment delayed the study for over a year. During this time, lab priorities and direction shifted and this study is no longer being conducted.
Sponsor: CommonSpirit Health (Other)
Collaborators: University of Colorado, Colorado Springs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1864889
Record Dates: First submitted 2022-07-26; First posted 2022-08-08 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2023-12

CONDITIONS: Body Temperature Changes; Exercise; Blood Pressure
MeSH Terms: conditions — Body Temperature Changes; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Does muscle temperature influence heat loss responses independently from core and skin temperature? (Experimental): The study will consist of three experimental trials, conducted in a randomized order, where participants will be required to run for one hour at ~60% of their maximal oxygen consumption on one of three different inclines: 1) flatland, 2) uphill, and 3) downhill. Environmental conditions will be maintained at 34°C/93°F and 20% relative humidity.
  Interventions: Procedure: Uphill running; Procedure: Flatland running; Procedure: Downhill running
- Does muscle temperature influence muscle blood flow independently from core and skin temperature? (Experimental): Following the exercise protocol described above in Arm 1, the participants will then lay supine for one hour while their muscle and skin blood flow, as well as blood pressure are measured.
  Interventions: Procedure: Uphill running; Procedure: Flatland running; Procedure: Downhill running
- What factors contribute to exercise-induced skeletal muscle damage? (Experimental): For those participants who additionally agree to participate in the muscle microdamage portion of the study, participants will be asked to return to the lab 24h and 48h post-trial. During these subsequent follow-up sessions, an additional blood sample will be drawn from the participants, the participants maximal voluntary contraction and muscle pain will be assessed, and they will be asked to fill out the muscle soreness scale.
  Interventions: Procedure: Uphill running; Procedure: Flatland running; Procedure: Downhill running

INTERVENTIONS:
Procedure: Uphill running — Participants will run at 70% of their maximal oxygen consumption for 60 min at a 10 degree (17.6%) incline.
Procedure: Flatland running — Participants will run at 70% of their maximal oxygen consumption for 60 min at a 0 degree (0%) incline.
Procedure: Downhill running — Participants will run at 70% of their maximal oxygen consumption for 60 min at a -10 degree (-17.6%) decline.

SUMMARY:
In animal models of thermoregulation (how the body regulates heat), heat-sensitive nerve cells that help regulate body temperature have been identified throughout the body (e.g. in muscles, viscera, and blood vessels, among others); however, in human thermoregulation models, only two locations are generally recognized: the core (brain) and the skin. The limited number of recognized locations in humans are likely due to the difficulty in testing these locations in humans, as these locations are typically identified in animals by sedating them, surgically opening them up, stimulating the area of interest with a hot or cold probe, and then measure thermoregulatory responses.

Based on the literature, the researchers believe that by having participants run at the same energy expenditure but at three different inclines (uphill, downhill and flat) on a treadmill, the researchers can independently alter muscle temperature, while keeping core and skin temperature the same. Additionally, recent studies have suggested that temperature has a greater role at regulating blood flow through muscle tissue than previously recognized. Because of this, the researchers aim to have a second arm of the study to see whether these differences in muscle temperature result in differences in post-exercise blood flow to the muscle.

Finally, downhill running is often used to study exercise-induced muscle damage, due to the greater breaking forces compared to flat land running. Because of this, a third study aim will be to examine the association between fitness level, body morphology and sex on exercise-induced muscle damage.

DETAILED DESCRIPTION:
Primary aim: To alter muscle temperature independently from core and skin temperature, to investigate the existence of temperature sensitive nerve cells in human muscle tissue.

In animal models of thermoregulatory control, multiple loci of thermal sensation have been identified, including in the muscle, veins in the skin and abdomen, spinal column, upper airway, abdominal wall, lower esophagus, stomach, and small intestine. In contrast to these animal models, in human models of thermoregulatory control, typically, only thermal inputs from the brain (usually represented as "core" temperature, with proxy measures taken at the esophagus, rectum, intestine, or aural canal) are considered, along with further inputs from the skin that modify the central brain signaling.

The limited number of recognized thermally sensitive locations in humans are likely not due to a truly small number of thermally sensitive loci, but rather, due to the difficulty in testing these locations in humans. Indeed, the typical model for identifying thermally sensitive locations in animals is to sedate them, surgically open them up, stimulate the area of interest with a hot or cold probe, and then measure thermoregulatory responses; a protocol that is clearly unacceptable in humans.

Supporting the idea that the lack of recognized thermally sensitive locations is due to testing limitations, rather than an actual non-existence of physical locations, the principal researcher on the current application (Dr. Morris) previously conducted a series of studies providing evidence for the existence of thermoreceptors in the human abdomen. Indeed, recent reviews regarding human thermoregulatory control have updated the number of thermally sensitive sites to include the abdomen.

In the present study proposal, the investigators believe to have identified a protocol which would identify another thermally-sensitive location: human skeletal muscle.

The method for measuring heat balance in humans can be expressed using the following equation:

M ± W = K ± C ± R + E

Where M is metabolic energy expenditure, W is the amount of energy exchanged with the environment via mechanical work, K is conduction, C is convection, R is radiation and E is evaporation. Here, if M ± W exceeds K ± C ± R + E, there will be heat storage in the body and core temperatures will rise. Conversely, if K ± C ± R + E exceeds M ± W, there will be a net heat loss from the body and core temperatures will decrease. However, as humans are homeotherms, the body will typically regulate itself so that both sides of the equation are equal. With heat stress, this is primarily done through an increase in sweating that increases evaporative heat loss.

From the above, this would indicate that if the external work is manipulated while metabolic energy expenditure is kept constant, a proportional, inverse change on the heat loss side of the equation (primarily through evaporation) is required. One way to manipulate external work is by running at different inclines and declines, as the amount of external work performed during running can be calculated as the vertical displacement of the individual, multiplied by their mass and acceleration due to gravity.

This type of study protocol has only been employed twice: both times in the 1960s and both using only three male participants. In the first study, it was observed that when running uphill compared to flatland, evaporative heat loss was lower (due to decreased sweating) by the exact amount of energy as calculated to how much was lost to the environment via external work (as would be predicted). Of note, however, was that core and skin temperature - the two recognized thermally sensitive areas in humans - were similar between both trials. Similarly, in the second study, when running uphill compared to flatland, evaporative heat loss decreased (consequent of decreased sweating) proportionally to the amount of heat lost to external work from running uphill. Also, when running downhill compared to running uphill, the evaporative heat loss increased (due to increased sweating) in proportion to the amount of heat that the was gained from the environment from running downhill. Again, core and skin temperature were similar in all three trials.

The change in evaporative heat loss (consequent of changes in sweating) combined with the lack of difference in core and skin temperature in both studies suggests the existence of thermoreceptors in a bodily location other than the core and skin. The most likely area being the muscles of the leg, as was noted by the author in the second study. The reason for this can be explained accordingly:

Imagine riding a bicycle. The energy needed to get a person moving is produced within the body, however, the energy to slow a person down is produced by activating their brakes, which causes friction between the brakes and their tires and the tires and the road. If a person were to touch their brakes and tires after applying the brakes, both tires and brakes would feel hot due to the friction used to slow the person down. Humans do not have external brakes like bicycles, but instead, rely on their legs to do both the accelerating and braking. As more work needs to be done to overcome gravity while going uphill compared to flatland running, the horizontal component (i.e. horizontal running speed) will be slower when running at an equivalent metabolic energy expenditure. Conversely, when running downhill compared to flatland, the body is being "helped" by gravity, and therefore, to maintain an equivalent energy expenditure, the person needs to run faster. Accordingly, more braking actions occur in the legs while running downhill, resulting in more frictional braking and therefore more heat stored locally within the muscle. This, however, has yet to be confirmed empirically.

Of importance, the two previously conducted studies in which external work was manipulated while metabolic energy expenditure was kept constant included exclusively male participants. Women (at least when tested during the early to mid-follicular phases of the menstrual cycle) appear to have lower end-exercise core and skin temperatures, but higher active/inactive skeletal muscle temperatures, compared to males following exercise. Additionally, mechanisms for whole body evaporative heat loss are attenuated in females compared to males due to a lower sweat gland output and sweat rate. This sex-difference effect seems to become larger in endurance trained versus untrained populations. As such, it is plausible that in situations which demand greater evaporative heat loss to accommodate for more heat stored locally in the skeletal muscle (i.e., downhill running), females will demonstrate a greater increase in muscle temperature relative to flatland running due to an inability to increase sweat rate beyond a certain threshold.

Therefore, if the hypotheses of this study are proved correct, the results from this study would demonstrate that humans have thermoreceptors residing in areas of the body, other than the core and skin, that can affect whole-body heat loss responses. In addition to providing fundamental knowledge about how the human body thermoregulates, these results could affect policies in place regarding whole-body warming and cooling protocols used in emergency, athletic, and surgical scenarios. Furthermore, given the limited amount of thermoregulatory research that has included women, successful completion of this study could influence sex-specific practices for thermal safety.

Secondary aim: Investigate whether muscle temperature influences muscle blood flow, and consequently, post-exercise hypotension.

In addition to answering questions regarding thermoregulatory control, the present study-design's ability to independently alter muscle temperature from skin and core temperature can be used to answer question regarding the effect of local muscle temperature on blood flow. Elevated muscle temperature has been associated with changes in cardiovascular control and greater post exercise vasodilation in the previously active muscle. However, muscle is typically heated externally, which concomitantly alters skin temperature, which also has major effects on local and skin blood flow. Accordingly, the present methodology will allow us to alter muscle temperature while keeping core and skin temperature consistent between trials, allowing us to study the independent effect of muscle temperature on muscle blood flow. Moreover, the investigators believe this will be the first attempt to compare the effects of muscle temperature mediated differences in muscle blood flow between men and women.

Tertiary aim: Downhill running, of similar duration and intensity to the proposed downhill trial in this study (i.e. 60% of maximum oxygen uptake [VO2max], on a -10% decline, for 60 min), is regularly used to study exercise-induced muscle damage. Specifically, previous studies have employed men running for 40 min at 70% VO2max on a -10% decline, 30 min at 70% VO2max on a -15% decline, 60 min at 65% VO2max on a -10% decline, 60 min at 65% VO2max on a -10% decline, and women running for 60 min at 75% VO2max on a -10% decline. Of particular note, although downhill running-induced muscle damage has been studied in men and women, only one within-study sex comparison has been performed. In this study, where participants ran for 30 min at 70% of their VO2max on a -15% incline, it was observed that male participants had higher markers of exercise-induced muscle damage, compared to the female group, 24 h post-exercise. Also, of note, no studies to date have looked at the interactions between sex and incline (i.e. downhill vs flatland vs uphill) on muscle damage. Therefore, the investigators intend to take measures of muscle damage as the investigators are performing these incline running trials anyway.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be healthy with no history of respiratory, metabolic, cardiovascular, blood pressure disease, or of diabetes and must not currently be on any medication related to these or any other conditions. Additionally, due to the potential dangers of elevated body temperatures to the unborn fetus, all female participants must not be pregnant and agree to not to attempt to become pregnant throughout their involvement in the study.

Exclusion Criteria:

* Unhealthy, history of respiratory, metabolic, cardiovascular, blood pressure disease, or of diabetes, currently taking medications related to these or that have the possibility of impairing cardiovascular or thermoregulatory function. Any participants that are pregnant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Core temperature | Immediately after completing the intervention
  Measured by rectal and esophageal temperature
Skin temperature | Immediately after completing the intervention
  Measured at 8 sites using the ISO 9886 weighting system
Muscle temperature | Immediately after completing the intervention
  Measured at 4 locations: vastus lateralis, bicep femoris, lateral gastrocnemius and deltoid
Whole-body sweat rate (arm 1) | Immediately after completing the intervention
  Measured pre and post exercise with a platform scale (accurate to 1 g)
Femoral blood flow (arm 2) | 1 hour after completing the intervention
  Measured using Ultrasound Doppler
Blood pressure (arm 2) | 1 hour after completing the intervention
  Measured using a standard blood pressure cuff and finger photoplethysmography
Perceived muscle pain (arm 3) | Assessed 48 hours after the completing exercise
  Self-reported on a 100 mm likert scale ranging from "no pain or discomfort" to "maximal pain and discomfort"
Maximal voluntary contraction (arm 3) | Assessed 48 hours after the completing exercise
  The maximal force (in N) generated by the right leg during an isometric leg extension, with the knee at 90 degrees
Plasma creatinine levels (arm 3) | Assessed 48 hours after the completing exercise
  Measured from blood taken from an ante cubital vein

SECONDARY OUTCOMES:
Oxygen consumption | Average oxygen consumption over the 60 min of exercise
  Measured by expired gas analysis an expressed as liters per minute
Local sweat rate | Average local sweat rate over the 60 min of exercise
  Measured using the ventilated sweat capsule technic
Skin blood flow | Average skin blood flow over the 60 min of exercise
  Measured using laser doppler
Heart rate | Average heart rate over the 60 min of exercise
  Using 3-lead ECG
Perceived exertion | Average perceived exertion over the 60 min of exercise
  Using the standard 15-point Borg Scale of perceived exertion ranging from no exertion (6) to extremely hard (20)
Thermal comfort | Average thermal comfort over the 60 min of exercise
  Using the Kansas State University 9-point thermal comfort model ranging from very cold (-4) to very hot (4)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan B Morris, PhD, Principal Investigator — University of Colorado, Colorado Springs

IPD SHARING:
Plan to Share IPD: Yes
Upon the completion of the study, a permanent link will be created to the data summary sheet containing the participants' deidentified data, as it was entered in the statistical software program used for the final analysis (Graphpad Prism or SPSS).
Time Frame: Data will be posted upon completion of the study, when the manuscripts are submitted for publication. This data will be available at the provided link for the foreseeable future.
Access Criteria: Open to all.